CLINICAL TRIAL: NCT03402490
Title: Enhancement of Physical Activity in Elderly Patients With Diastolic Heart Failure by a Motivational Intervention - Pilot Data From an add-on Following the Ex-DHF Trial
Brief Title: Enhancement of Physical Activity in Elderly Patients With Diastolic Heart Failure by a Motivational Intervention
Acronym: Ex-DHFadd-on
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Göttingen (Other)
Collaborators: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other)
Responsible Party: Principal Investigator, Christoph Herrmann-Lingen, Prof. Dr., University of Göttingen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 12345 add-on
Record Dates: First submitted 2017-12-22; First posted 2018-01-18 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Diastolic Heart Failure
Keywords: Motivational interviewing; physical activity; feasibility; HFpEF
MeSH Terms: conditions — Heart Failure, Diastolic; Motor Activity | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: One group of participants received motivational counseling to enhance physical activity; the other group received usual care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational interviewing (Experimental): Over a time span of 6 months, participants in the intervention group received up to 7 sessions of motivational counseling, lasting 15-30 minutes each, to enhance physical activity.
  Interventions: Behavioral: Motivational interviewing
- Usual care (No Intervention): Participants who served as controls received usual care.

INTERVENTIONS:
Behavioral: Motivational interviewing
  Arms: Motivational interviewing

SUMMARY:
The aim of our pilot study is to evaluate the feasibility, acceptance and efficacy of motivational interviewing (MI) to support elderly patients with heart failure with preserved ejection fraction (HFpEF) in maintaining or starting physical activity (PA).

DETAILED DESCRIPTION:
Patients discharged from the Ex-DHF trial were recruited from June 2013 to December 2015 and offered participation in a controlled add-on pilot study. The treatment group (n=19) received 5 sessions of MI, each lasting 15-30 min over 6 months to enhance physical activity.

For the first two and the last sessions participants met with the psychologist-counsellor face-to-face for about 45 minutes. The remaining three sessions could be conducted via telephone or face-to-face, depending on participants' preferences, and typically lasted 15-30 minutes. Per study protocol, counsellors (physicians and psychologists trained in motivational interviewing) assisted the participants in: (1) Setting goals for their physical activity; (2) developing a plan to increase physical activities; (3) setting specific plans for the implementation of the plan; and (4) overcoming possible barriers. Participants were also asked to keep track of their daily physical activity in a diary, which counsellors then discussed with them during the sessions.

After patients had given their written informed consent, counsellors assessed all participants via structured interview and self-rating scales. At baseline only, sociodemographic information was recorded.

At baseline and at the final 6-month visit participants' motivation to be physically active in the upcoming weeks was assessed using the SSK-scale ("Sportbezogene Selbstkonkord" = sports-related self-concordance, Seelig and Fuchs 2006) to assess the self concordance of sport- and exercise-related goals.

The kind and extent of patients' daily physical activity was recorded using patient diaries. At baseline and 6 months we also conducted a symptom-limited cardiopulmonary exercise test on a bicycle ergometer, in order to assess changes in maximum rate of oxygen consumption during the last 30 seconds before the termination of the exercise (peak oxygen consumption (VO2 [ml/min/kg])) as measure of maximal exercise capacity. Participants also completed the 6-minute walk test on flat surface (6-MWT) as an additional parameter to assess submaximal exercise capacity.

Additionally, at the 6-month assessment, intervention participants filled out a questionnaire about their subjective evaluation of the counseling program.

The control group (n=20) received usual care.

ELIGIBILITY:
Inclusion Criteria:

* preserved left ventricular systolic function (left ventricular ejection fraction >= 50%),
* echocardiographically determined diastolic dysfunction (grade ≥ 1),
* New York Heart association functional classes I, II or III,
* at least one cardiovascular risk-factor (overweight, diabetes, hypertension, smoking or hyperlipidemia)
* participation in Ex-DHF main study
* written informed consent

Exclusion Criteria:

* Non-cardiac causes for heart failure-like symptoms
* Chronic obstructive pulmonary disease GOLD stages ≥II
* Anaemia (haemoglobin <11 mg/dL)
* Significant renal dysfunction (eGFR <30 mL/min/1.73 m**2 indexed to BSA)
* Significant peripheral artery disease (Fontaine ≥IIb)
* Musculoskeletal disease that contributes to reduced exercise performance
* Specific cardiomyopathy (e.g. amyloidosis)
* Haemodynamically significant valvular disorders
* Significant coronary artery disease (current angina pectoris Canadian Cardiovascular Society Class ≥II or positive stress test, myocardial infarction or coronary artery bypass graft within the last 3 months)
* Any inability or contraindication to participate in cardiopulmonary exercise testing or in an exercise programme (e.g. physiological, mental) or to supply essential information (e.g. questionnaire, diary)
* Ineffective control of resting blood pressure (≥140/90 mmHg or ≥160/100 mmHg with ≥3 antihypertensive drugs) or of resting heart rate (≥100 b.p.m.)
* Expected low adherence (e.g. by travel distance to trial site; planned absences longer than 4 weeks during follow-up) or ongoing drug abuse
* Pregnant or nursing women
* Concomitant participation in other interventional clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-06-18 (Actual); Primary Completion 2015-12-08 (Actual); Study Completion 2015-12-08 (Actual)

PRIMARY OUTCOMES:
Adherence to intervention | Over 6 month intervention period
  To evaluate the feasibility of motivational counseling to enhance physical activity patients´ adherence to appointments is assessed as number / percentage of sessions attended
Patient acceptance of intervention | At 6-month assessment
  To assess how patients evaluate the Intervention, i.e. receiving motivational counseling, they were asked to fill in evaluation sheets
Effectiveness (peak VO2) | Change from baseline to 6-month assessment
  Changes in the maximal exercise capacity (peak VO2) during a symptom-limited cardiopulmonary exercise test on a bicycle ergometer.
Effectiveness (6-minute walk distance) | Change from baseline to 6-month assessment
  Six-minutes walking distance

OTHER OUTCOMES:
Motivation | Change from baseline to 6-month assessment.
  Participants' motivation to be physically active was registered using the SSK (Sports-related self-concordance) scale. The self-concordance score is computed by subtracting the sum of the introjected and extrinsic motivation from the sum of the intrinsic and identified motivation subscales, with resulting scores ranging from -10 to +10 (higher value = higher self-concordance)
Physical activity | Change from baseline to 6-month assessment.
  The kind and extent of patients' daily physical activity was recorded using patient diaries